CLINICAL TRIAL: NCT00396500
Title: To Assess the Effectiveness of Six-Monthly Deworming With Vitamin A Administration on Growth in 1-5 Year Old Children in the Urban Slums of Lucknow
Brief Title: Deworming and Vitamin A (DEVTA) Prepilot Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: King George's Medical University (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 01
Record Dates: First submitted 2006-11-04; First posted 2006-11-07 (Estimated); Last update posted 2006-11-07 (Estimated); Status verified 2006-11

CONDITIONS: Malnutrition; Worm Infestation; Under-Fives
Keywords: Deworming; Malnutrition; children; Community; India
MeSH Terms: conditions — Malnutrition; Trematode Infections | interventions — Albendazole; Vitamin A

INTERVENTIONS:
Drug: Albendazole (400 mg) and/or Vitamin a

SUMMARY:
Background. More than a third of the world's population is infected with intestinal nematodes. A majority of these infections occur in children. Current control approaches emphasise treatment of school age children, and there is a lack of information on the effects of deworming preschool childrenSetting: Within the Integrated Child Development System (ICDS) infrastructure in urban Lucknow (UP), IndiaDesign: Open Labeled randomised trialHypothesis: Our study hypothesis was that albendazole administration six monthly, as a single 400 mg dose in syrup, by the existing health care delivery system would be a practicable way to achieve mass deworming of preschool children and this might result in an improvement in weight gain of preschool childrenIntervention One group will receive usual health care by the existing health care staff, which included six monthly administration of Vitamin A concentrate. The other group will receive, in addition, 400 mg of albendazole (Zentel, Smith Kline & Beecham) in 10 ml syrup form. Five such doses will be given at six monthly intervals for 2 years.Main objective: To assess the impact of 6 monthly deworming on weight and height gain at the end of 2 years in children aged 1 to 5 years of age Main outcomes measures: Weight gain in 2 yearsInclusion criteria: Children 1 to 5 years, whose guardians give written informed consent. Exclusion criteria: Those not consentingSample size: Sample size was calculated for a continuous outcome. For a standardized effect size of 0.1, with a power of 80% and an alpha level of 0.05, using a 2-tailed t test, taking into account design effect, about 2000 children will be included in each arm.

ELIGIBILITY:
Inclusion Criteria:

* Local residents
* Aged 1-5 years
* Informed written parental consent

Exclusion Criteria:

* Refusal to give consent
* prior enrollment in the study

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4000
Dates: Start 1994-04; Study Completion 1996-12

PRIMARY OUTCOMES:
Change in weight in 2 years

SECONDARY OUTCOMES:
Secondary: Weight and Height gain in underweight, stunted and wasted children

CONTACTS AND LOCATIONS:
Overall Officials: Shally Awasthi, MD, DNB, Principal Investigator — Dept of Pediatrics, King George's Medical University, Lucknow, India
Locations (1):
- Lucknow Commission, Lucknow, Uttar Pradesh, India

REFERENCES:
- [Derived] Awasthi S, Peto R, Pande VK, Fletcher RH, Read S, Bundy DA. Effects of deworming on malnourished preschool children in India: an open-labelled, cluster-randomized trial. PLoS Negl Trop Dis. 2008 Apr 16;2(4):e223. doi: 10.1371/journal.pntd.0000223. PMID 18414647